CLINICAL TRIAL: NCT04652115
Title: A Single-Arm Safety and Feasibility Study of Defibrotide for the Treatment of Severe COVID-19
Brief Title: Defibrotide for the Treatment of Severe COVID-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Paul G. Richardson, M.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P003203
Record Dates: First submitted 2020-12-01; First posted 2020-12-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — defibrotide

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, two cohort clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Defibrotide (Experimental): Defibrotide IV
  Interventions: Drug: Defibrotide

INTERVENTIONS:
Drug: Defibrotide — Deibrotide via IV

SUMMARY:
The goal of this study is to evaluate the safety and feasibility of defibrotide in COVID-19 pneumonia.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, two-cohort, phase 2 pilot study that will evaluate the safety and efficacy of defibrotide in clinically severe COVID-19. The defibrotide dose that is approved by the FDA for the treatment of post-HSCT VOD/SOS (6.25 mg/kg IV q6 hours) will be used.

Cohort 1 will consist of patients with COVID-19 pneumonia confirmed by PCR and radiography, who are hospitalized with an oxygen requirement (either supplemental O2 or mechanical ventilation), are not on therapeutic dose anticoagulation, and require no more than one vasopressive agent to maintain hemodynamic stability. Cohort 2 will consist of patients with COVID-19 pneumonia confirmed by PCR and radiography, who are hospitalized in the ICU and are at elevated risk of hemorrhage and/or hypotension, the former defined as a requirement for therapeutic dose anticoagulation for active thrombosis, ECMO, or CRRT, and the latter defined as a requirement for two vasopressive agents to maintain hemodynamic stability.

In cohort 2 only, a 6+6 dose de-escalation design will be utilized, in which if 2 of 6 DLTs are experienced in the first 6 subjects, the dose will be reduced from 6.25 mg/kg IV q6hrs to 10mg/kg/d CIVI. If there are 0 or 1 DLTs in the first 6 subjects at the FDA-approved dose, another 6 subjects will be enrolled at the same dose. Grade 3/4 hemorrhage and significant new hypotension will be considered DLT's.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Active COVID-19 infection confirmed by positive SARS-CoV-2 PCR.
3. Radiographic evidence of bilateral pulmonary infiltrates.
4. A life expectancy of at least 24 hours.
5. Score of 4-7 on the WHO ordinal scale.
6. Prophylactic dose anticoagulation is allowed for enrollment into cohort 1. Therapeutic dose anticoagulation for active thrombosis, ECMO, and/or continuous renal replacement therapy (CRRT) is allowed for enrollment into cohort 2 if there is no evidence of bleeding after at least 24 hours of anticoagulation.
7. Patient or surrogate able to provide informed consent

Exclusion Criteria:

1. Clinically significant acute bleeding.
2. Concomitant use of thrombolytic therapy (e.g. t-PA).
3. Hemodynamic instability, defined as a requirement for >1 vasopressor agent for enrollment into cohort 1, and a requirement for >2 vasopressor agents for enrollment into cohort 2
4. Known allergy or hypersensitivity to DF.
5. Pregnant or lactating.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse event of special interest (bleeding and hypotension) | Up to 21 days
  The rate of adverse event of special interest (bleeding and hypotension)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States